CLINICAL TRIAL: NCT05115643
Title: Examining Changes in Muscle Size and Strength, Neuromuscular Function, and Brain Plasticity During Limb Immobilization in Women
Brief Title: Brain and Muscle Plasticity During Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Assistant Professor, McGill University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A00-M01-21A
Record Dates: First submitted 2021-10-10; First posted 2021-11-10 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Immobilization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilized arm (Experimental): Left arm of participant
  Interventions: Behavioral: Immobilization
- Non-immobilized arm (No Intervention): Right arm of participant

INTERVENTIONS:
Behavioral: Immobilization — Immobilization of left arm using a brace and sling.
  Arms: Immobilized arm

SUMMARY:
Patients in rehabilitation may undergo periods of prolonged limb immobilization in response to injury, surgery, or illness. Due to disuse, the size and strength of muscles controlling the affected limb can decrease significantly, possibly resulting in physical impairment or lower quality of life during the recovery phase. Prior immobilization studies have shown that the rate and degree of decline in muscle strength exceeds that of muscle size, indicating that determinants of muscle strength unrelated to muscle size may further contribute to functional changes during immobilization.

The purpose of this study is to describe the changes in muscle strength, muscle size, corticospinal excitability, voluntary activation, M1 cortical thickness, and resting state functional connectivity following a 2-week limb immobilization period in young women.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female
* Right-hand dominant
* Body mass index between 18.5-30 kg/m^2 (inclusive)
* Regular menstrual cycle
* Be able to maintain a habitual diet throughout the duration of the study

Exclusion Criteria:

* Use of tobacco
* Pregnancy
* A history of brain trauma
* Suffers from a neurological disease or movement disorder
* Peripheral nerve damage
* Use of medications known to affect protein metabolism (i.e., corticosteroids, non-steroidal anti-inflammatory drugs, or prescription strength acne medications)
* Diagnosed with or suspects having a psychiatric illness
* Use of dietary supplements known to affect muscle size (i.e., creatine, fish oil)
* Past or present diagnosis of an eating disorder by a physician or registered dietician
* Possesses any metal implants (e.g. artificial joints, pacemakers, stents) or non-removeable medical devices that are contraindicative for magnetic resonance imaging (e.g. insulin pumps)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Change in isometric elbow flexion and extension peak torque, both arms | Comparison between before and after 2 weeks of left arm immobilization
  Measured using an isokinetic dynamometer; peak torque during static contraction of the elbow flexors and extensors
Change in isokinetic elbow flexion and extension peak torque, both arms | Comparison between before and after 2 weeks of left arm immobilization
  Measured using an isokinetic dynamometer; peak torque during dynamic contraction of the elbow flexors and extensors
Change in cross-sectional area of the elbow flexor and extensor muscles, both arms | Comparison between before and after 2 weeks of left arm immobilization
  Obtained from magnetic resonance images of each arm
Change in volume of the elbow flexor and extensor muscles, both arms | Comparison between before and after 2 weeks of left arm immobilization
  Obtained from magnetic resonance images of each arm
Voluntary activation of biceps brachii, both arms | Comparison between before and after 2 weeks of left arm immobilization
  Measured using peripheral nerve stimulation and an isokinetic dynamometer; estimation of the capacity to voluntarily activate the force-generating elements of the biceps brachii during maximal effort elbow flexion
Change in corticospinal excitability of biceps brachii, both arms | Comparison between before immobilization and 24 hours of left arm immobilization, and before and after 2 weeks of left arm immobilization
  Measured using transcranial magnetic stimulation; estimation of the efficacy of the corticospinal tract to relay electrical signals to the biceps brachii muscle

SECONDARY OUTCOMES:
Change in right and left primary motor cortex thickness | Comparison between before and after 2 weeks of left arm immobilization
  Obtained from magnetic resonance image of the brain
Change in whole brain resting state functional connectivity | Comparison between before and after 2 weeks of left arm immobilization
  Obtained from magnetic resonance image of the brain

OTHER OUTCOMES:
2-day caloric and macronutrient intake, before immobilization | Measured during the 2-day period right before left arm immobilization
  Obtained using self-reported dietary intake records
2-day caloric and macronutrient intake, during immobilization | Measured during the last 2 days of left arm immobilization
  Obtained using self-reported dietary intake records
Ovarian hormone concentrations (estradiol, progesterone) | Measured on day of left arm immobilization, before putting on the arm brace
  Obtained using blood samples
Ovarian hormone concentrations (estradiol, progesterone) | Measured after 2 weeks of left arm immobilization
  Obtained using blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism and Nutrition Research Laboratory, Montreal, Quebec, Canada